CLINICAL TRIAL: NCT05085522
Title: Study of the Effect of Systematic Screening of Residents and Caregivers by Nasopharyngeal Swab (RT-PCR) on the Incidence Rate of COVID-19 Infection in Medico-social Institutions for the Elderly
Brief Title: Study of the Effect of Systematic Screening of Residents and Caregivers With Covid-19 by Nasopharyngeal Swab (RT-PCR)
Acronym: INMESO-Covid
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7953
Record Dates: First submitted 2021-10-07; First posted 2021-10-20 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-10

CONDITIONS: COVID-19
Keywords: COVID-19; RT-PCR; SARS-CoV-2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The current COVID-19 epidemic has overwhelmed the health systems of many countries in which it has broken out, forcing various governments to institute population containment measures.

Residents of medico-social institutions for the elderly are particularly at risk of developing severe forms because they have a large number of factors favoring the progression to a severe form (very advanced age, multiple comorbidities, dependence in activities of dayli life).

The specificity and positive predictive value of clinical signs are not very important in this population; which makes the diagnosis even more complicated.

One of the strategies to try to protect these residents, in addition to room containment and clinical surveillance, would be to carry out a systematic screening campaign of all residents and all caregivers, then to consider reorganizing the establishments with a sector "COVID +".

This was announced by the French Minister of Health Olivier VERAN on 04/06/2020 from the first confirmed case of COVID-19 in an institution.

However, asymptomatic subjects may have a "negative" RT-PCR test at one point but which is positive in the following days. And in this interval they would still be contagious.

It is therefore not excluded that the implementation of such a screening campaign will not be effective in reducing the number of new cases of COVID-19 in medico-social institutions for the elderly

ELIGIBILITY:
Inclusion criteria:

* Major subject (≥18 years old)
* Subject hospitalized in a medico-social institution for the elderly (SMTI or EHPAD) at the HUS or in another center which will be recruited secondarily and whose patients in a unit all have the same attending physician.
* Subject (or family) who did not express their disagreement with the reuse of this data for the purposes of this research.

Exclusion criteria:

* Subject having expressed opposition to participating in the study
* Subject under guardianship or guardianship
* Subject under safeguard of justice

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Major subject (≥18 years old) hospitalized in a medico-social institution for the elderly (SMTI or EHPAD) at the HUS or in another center which will be recruited secondarily and whose patients in a unit all have the same attending physician.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-01-30 (Estimated); Study Completion 2022-01-30 (Estimated)

PRIMARY OUTCOMES:
Retrospective study of the effect of systematic screening of residents and caregivers by nasopharyngeal swab (RT-PCR) on the incidence rate of COVID-19 infection | Files analysed retrospectively from March 15, 2020 to July 31, 2020 will be examined]

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre BOUSSUGE, MD, Principal Investigator — Service Gériatrie. Soins Médico-techniques Importants - Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service Gériatrie. Soins Médico-techniques Importants - Hôpitaux Universitaires de Strasbourg, Strasbourg, France